CLINICAL TRIAL: NCT06111716
Title: The Effect of Mindfulness-Based Childbirth Education on Psychosocial Outcomes in Pregnant Women: A Randomized Controlled Study
Brief Title: Mindfulness in Childbirth Preparation Education Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Sibel OCAK AKTURK, Principal Investigator, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PhDThesis
Record Dates: First submitted 2023-10-21; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Pregnant Women
Keywords: Mindfulness; Depression; Pregnant Women; Childbirth Education; Self-efficacy; Postpartum trauma
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Mindfulness-Based Childbirth Education was implemented in the intervention group
  Information-Based Birth Education was applied to the control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information-Based Childbirth Education Group (Active Comparator): Information-Based Birth Preparation Education Content; "Physical and mental preparation for birth, the birth process, non-pharmacological methods that reduce birth pain and facilitate birth, postpartum period characteristics, physiological and psychological effects on the mother after birth."It includes topics such as "changes, adaptation to the maternal role, newborn care". Education is information-based, not based on a philosophy or model.
  Interventions: Other: Information-Based Birth Education
- Mindfulness-Based Childbirth Education Group (Experimental): Mindfulness-Based Childbirth Education includes topics related to birth as well as mindfulness, mindfulness attitudes and practices, mindfulness in daily life, mindfulness during pregnancy and postpartum period, mindfulness breastfeeding and meditation practices. The training duration is 8 weeks (2 hours each week).
  Interventions: Other: Mindfulness- Based Childbirth Education

INTERVENTIONS:
Other: Mindfulness- Based Childbirth Education — Mindfulness- Based Childbirth Education Group includes; Women were given eight-week birth preparation training. In this training, in addition to information about birth, mindfulness, mindfulness attitudes and practices, mindfulness in daily life, mindfulness in pregnancy and postpartum period, mindfulness breastfeeding and meditation practices were included.
  Arms: Mindfulness-Based Childbirth Education Group
Other: Information-Based Birth Education — In the Information-Based Birth Education Group, women were given 4-week (4 hours per week) birth preparation training. The education given was not based on a philosophy or method.
  Arms: Information-Based Childbirth Education Group

SUMMARY:
The study was conducted as a prospective, randomized controlled study to determine the effect of Mindfulness-Based Childbirth Education on psychosocial outcomes in pregnant women. Pregnant women applied to Istanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Department of Obstetrics and Gynecology, Pregnancy Polyclinic and Faculty Member Polyclinic between 15.09.2021-28.06.2022. A total of 82 pregnant women were included in the experimental and control groups. The experimental group received Mindfulness-Based Childbirth Education for 8 weeks and the control group received Information-Based Childbirth Education for 4 weeks. Evaluation was performed in both groups before and after the training and at the end of the 4th postpartum week. The data were collected using the Introductory Information Form, Perceived Stress Scale, Edinburg Postpartum Depression Scale, Birth Self-Efficacy Scale and City Birth Trauma Scale.

DETAILED DESCRIPTION:
This prospective, randomized controlled study was conducted to determine the effect of Mindfulness-Based Childbirth Education on psychosocial outcomes in pregnant women. In this randomized controlled intervention study, the "Consolidated Standards for Reporting Studies (CONSORT) 2018" guideline was followed. It was conducted with pregnant women who applied to Istanbul University-Cerrahpaşa, Cerrahpaşa Medical Faculty using Zoom program, a web-based application. Faculty of Medicine, Department of Obstetrics and Gynecology, Pregnancy Polyclinic and Faculty Member Polyclinic, between 15.09.2021-28.06.2022. A total of 82 pregnant women were included in the experimental and control groups.

Preliminary Preparation and Creation of Education Content: The primary researcher (SOA) who provided the training received a Certificate of Mindfulness and Childbirth Preparedness Trainer Training. In order to evaluate the suitability of the content and scope of the Mindfulness-Based Childbirth Education, which was prepared in line with the literature, to the training received by the researcher, the opinions of 4 experts working on mindfulness and childbirth preparation training were obtained. The content of the training was prepared in line with the feedback received from the experts. Eight sessions were carried out as a pilot application to four pregnant women in order to determine the suitability of the content of the Mindfulness-Based Childbirth Education Training, to plan the duration of the training and to determine the points that were not understood in the training. At the end of the pilot application, the training content was finalized. Pilot application data were not included in the study.

Group Formation: The groups were randomized into two groups by an independent researcher using the web-based randomization program randomizer.org. Pregnant women who met the inclusion criteria were assigned numbers according to the sequence numbers obtained using the randomization program.

Interventions:

Information-Based Childbirth Education: The content of Information-Based Childbirth Education includes topics such as "Physical and mental preparation for childbirth, the birth process, non-drug methods that reduce birth pain and facilitate birth, postpartum period characteristics, physiological and psychological changes in the mother after birth, adaptation to the role of motherhood. newborn care." Since the pregnant women were included in the study starting from the 20th week, pregnancy-related topics were not included in the training content. The training program is organized for four hours each week for four weeks. At least four pregnant women attended each session. It was completed on the alternative training day planned for pregnant women who could not attend. Participants were given homework assignments at the end of each session and asked to complete these assignments by the next training session. After the training, the postpartum women were reminded weekly via WhatsApp until the end of the fourth week after the birth of the baby.

Mindfulness-Based Childbirth Education: In addition to the topics covered in the Information-Based Childbirth Preparation Training, mindfulness, mindfulness attitudes, practices, mindfulness in daily life, pregnancy and postpartum period, mindful breastfeeding and meditation practices are included. It is recommended that Mindfulness-Based Childbirth Education should include nine sessions lasting three hours per week and one full day of rest, and the ninth session should be held as a "meeting" after delivery. However, in our study, the participation of pregnant women in the training program was taken into consideration and in order to prevent loss of participants, the trainings were implemented as 2.5 hours and one full retreat day every week for eight weeks, as in many practices. There are studies on this subject in the literature. Considering the participants' unavailability on training days, an alternative training day was planned once a week. In the study, a minimum of four and a maximum of nine people participated in group trainings. At the end of each training session, a meditation practice lasting approximately 20 minutes was performed. At the end of each session, participants were told how to perform informal mindfulness practices (mindful eating, drinking coffee, walking) at home and were asked to repeat the formal meditation practices taught until the next training session. After the training, postpartum women were reminded weekly until the end of the fourth postpartum week to perform the formal and informal meditation practices included in the training provided within the scope of the study.

Data Collection: The licensed Zoom program, a web-based application, was used to deliver the training. A separate WhatsApp group was created for both groups in the study. Before starting the Prenatal Preparation Training, the first part of the Introductory Information Form, Perceived Stress Scale, Birth Self-Efficacy Scale and Edinburg Postpartum Depression Scale was created with Google Forms and the link was sent to the WhatsApp groups. Pregnant women in the groups filled out the forms using this link. After the Preparation for Childbirth Training ended (at the end of the eighth week for the Intervention group and at the end of the fourth week for the Control group), the Perceived Stress Scale, the Self-Efficacy in Childbirth Scale, and the Edinburgh Postnatal Depression Scale, linked to Google Forms, were sent to the WhatsApp groups. Pregnant women in the groups filled in the forms using this link. In the fourth week after delivery, the second part of the Descriptive Information Form created with Google Forms and the link to the Perceived Stress Scale, Edinburgh Postnatal Depression Scale and City Birth Trauma Scale were sent to the WhatsApp groups. Postpartum women in the groups completed the forms using this link.

Data Collection Tools Introductory Information Form: The form prepared in line with the literature consists of two sections and a total of 28 questions. In the first part of the form, there are a total of 20 questions evaluating the socio-demographic characteristics of pregnant women (12), descriptive characteristics such as alcohol habits and physical activity status (6) and birth history (2). In the second part, there are 8 questions evaluating the characteristics of the postpartum period.

Perceived Stress Scale (PSS-14/PSS): The scale consists of a total of 14 items and evaluates individuals' stress perceptions against certain situations they encounter in their lives. The scale has a five-point Likert rating. The scale has two subscales called "perception of insufficient self-efficacy" and "perception of stress/discomfort". Items 4, 5, 6, 7, 9, 10, 13, which contain positive statements, are reverse scored. The lowest score that can be obtained from ASÖ-14 is 0 and the highest score is 56. An increase in the scores people get from the scale indicates that their perception of stress increases. In the original development study of the scale, the Cronbach's alpha coefficient of PSS-14 was found to be 0.84. In our study, the Cronbach's alpha coefficient of the scale was found to be 0.65.

Childbirth Self-Efficacy Scale (CBSEI): The 62-item scale developed by Lowe was later developed by Ip et al. (2008) and abbreviated it as the Short Form of the Labor Self-Efficacy Scale. The scale evaluates women's self-efficacy level regarding labor. The CBSEI Likert-type scale has two subscales, outcome and competence expectancy, each consisting of 16 items. The first 13 items in competence expectation are reverse scored. The minimum score to be obtained from each sub-dimension of the scale is 16 and the maximum score is 160. The minimum score to be obtained from the entire scale is 32, and the maximum total score is 320. Increasing scores on the scale indicate that pregnant women's self-efficacy levels in labor are high.

Edinburgh Postnatal Depression Scale (EPDS): The 4-point Likert-type scale consists of a total of 10 questions assessing the psychological state of the respondent in the last week. It evaluates the risk of depression during pregnancy and postpartum period, but is not a measurement tool that can diagnose depression on its own. The lowest score that can be obtained from EPDS is 0 and the highest score is 30. 7 items (3,5,6,7,8,9,10) in the scale are reverse scored. The cut-off point of the scale is 12, and women with a total scale score of more than 12 are considered to be in the "risk group" for depression.

City Birth Trauma Scale (CBSEI-C32): The four-point Likert-type scale consists of 29 items and five sub-dimensions. Sub-dimensions; re-experiencing, avoidance symptoms, negative cognitions and mood, hyperarousal and dissociative symptoms.CBSEI is used to evaluate the symptoms of Post-Traumatic Stress Disorder (PTSD) and is not a diagnostic tool. Levels 1-2 on the scale. substances stress, 3-7. Items describe symptoms of re-experiencing labor, items 8-9. items avoidance symptoms, 10-16. questions about negative cognitions and mental state symptoms, 17-22. Items assess symptoms of overstimulation. 3-22. In the items, people rate the questions asked about their last week as "never", "1 time", "2-4 times", "5 or more times". 3-22. The total score range for the items is 0-60. An increase in the score obtained from the scale means that post-traumatic stress symptoms are more common and reflects a greater risk for Post-Traumatic Stress Disorder (PTSD).

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Being primiparous
* To be at least primary school graduate,
* Not having a risky pregnancy,
* Being between 20-26 weeks of pregnancy,
* Those who volunteered to participate in the study,
* Having internet access and equipment (computer, smart phone, etc.).

Exclusion Criteria:

* Being multiparous
* To have taken yoga or mindfulness training during pregnancy or before,
* Pregnant women with communication problems (related to hearing, speaking and understanding),
* Receiving psychiatric treatment during pregnancy or postpartum period.
* Pregnant women who want to leave the study,
* Those who were diagnosed with risky pregnancy during the research (preeclampsia, threat of premature birth, etc.),
* Pregnant women who do not attend 70% of the education.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Perceived Stress | from the beginning of the study to the fourth week postpartum
  The perceived stress level of pregnant women before and after the training was evaluated. Perceived stress level was re-evaluated at the 4th week postpartum. "Perceived Stress Scale (PSS)" was used to evaluate the perceived stress level. Perceived Stress Scale consists of a total of 14 items and evaluates individuals' stress perceptions against certain situations they encounter in their lives. The scale has a five-point Likert rating. The scale has two subscales called "perception of insufficient self-efficacy" and "perception of stress/discomfort".The lowest score that can be obtained from PSS-14 is 0 and the highest score is 56. An increase in the scores people get from the scale indicates that their perception of stress increases.
Self-Efficacy in Labor | From the beginning of the study to the end of training and birth
  Self-efficacy levels of pregnant women were evaluated before and after the training. A total of 2 measurements were made. "Self-Efficacy in Childbirth Scale" was used to assess the level of self-efficacy. The Self-Efficacy in Childbirth Scale evaluates women's self-efficacy level regarding childbirth. The scale has two subscales. The minimum score that can be obtained from each subscale is 16 and the maximum score is 160. The minimum score that can be obtained from the whole scale is 32 and the maximum total score is 320. Higher scores obtained from the scale indicate that pregnant women have higher levels of self-efficacy for childbirth.
Edinburgh Postpartum Depression Incidence | From the beginning of the study (pre-training) to the fourth week postpartum.
  The depression symptoms of the pregnant women were evaluated 3 times in total, before, after and at the fourth week after delivery. Edinburgh Postpartum Depression Scale was used in the evaluation. Self-efficacy levels of pregnant women were evaluated before and after the training. A total of 2 measurements were made. The "Self-Efficacy in Childbirth Scale" was used to assess the level of self-efficacy. The Self-Efficacy in Childbirth Scale evaluates women's self-efficacy level regarding childbirth. The scale has two subscales. The minimum score that can be obtained from each subscale is 16 and the maximum score is 160. The minimum score that can be obtained from the whole scale is 32 and the maximum total score is 320. Higher scores obtained from the scale indicate that pregnant women have higher levels of self-efficacy for childbirth.
Symptoms of post traumatic stretch disorder | In the fourth week postpartum
  Postpartum posttraumatic stress disorder (PTSD) symptoms were assessed only at the fourth postpartum week using the City Birth Trauma Scale. The four-point Likert-type scale consists of 29 items and five subscales. The sub-dimensions are re-experiencing, avoidance symptoms, negative cognitions and mood, hyperarousal and dissociative symptoms. The City Birth Trauma Scale is used to assess symptoms of Posttraumatic Stress Disorder (PTSD) and is not a diagnostic tool. A higher score on the scale means that posttraumatic stress symptoms are more prevalent and reflects a greater risk for Posttraumatic Stress Disorder (PTSD).

CONTACTS AND LOCATIONS:
Overall Officials: sibel Ocak Akturk, Principal Investigator — Çanakkale Onsekiz Mart University
Locations (1):
- Çanakale Onsekiz Mart University, Çanakkale, Turkey (Türkiye)

REFERENCES:
- [Background] Duncan LG, Cohn MA, Chao MT, Cook JG, Riccobono J, Bardacke N. Benefits of preparing for childbirth with mindfulness training: a randomized controlled trial with active comparison. BMC Pregnancy Childbirth. 2017 May 12;17(1):140. doi: 10.1186/s12884-017-1319-3. PMID 28499376
- [Result] Lonnberg G, Jonas W, Unternaehrer E, Branstrom R, Nissen E, Niemi M. Effects of a mindfulness based childbirth and parenting program on pregnant women's perceived stress and risk of perinatal depression-Results from a randomized controlled trial. J Affect Disord. 2020 Feb 1;262:133-142. doi: 10.1016/j.jad.2019.10.048. Epub 2019 Oct 30. PMID 31733457
- [Result] Duncan LG, Bardacke N. Mindfulness-Based Childbirth and Parenting Education: Promoting Family Mindfulness During the Perinatal Period. J Child Fam Stud. 2010 Apr;19(2):190-202. doi: 10.1007/s10826-009-9313-7. Epub 2009 Oct 10. PMID 20339571
- [Result] Fisher C, Hauck Y, Bayes S, Byrne J. Participant experiences of mindfulness-based childbirth education: a qualitative study. BMC Pregnancy Childbirth. 2012 Nov 13;12:126. doi: 10.1186/1471-2393-12-126. PMID 23145970